CLINICAL TRIAL: NCT04720963
Title: Intranasal Remimazolam for Premedication in Pediatric Patients: a Double-blinded Randomized Clinical Trial
Brief Title: Intranasal Remimazolam for Premedication in Pediatric Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2020-03-114
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Sedative; Anxiety Disorder
Keywords: remimazolam
MeSH Terms: conditions — Anxiety Disorders | interventions — remimazolam; Injections; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group P (Placebo group) (Placebo Comparator): intranasal placebo about 30min before anesthesia induction
  Interventions: Other: Distilled water for injection
- group R (remimazolam group) (Experimental): intranasal remimazolam about 30min before anesthesia induction
  Interventions: Drug: Remimazolam
- group D (Dexmedetomine group) (Active Comparator): intranasal dexmedetomidine about 30min before anesthesia induction
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — intranasal remimazolam
  Arms: group R (remimazolam group)
Other: Distilled water for injection — intranasal distilled water for injection
  Arms: group P (Placebo group)
Drug: Dexmedetomidine — Intranasal dexmedetomidine
  Arms: group D (Dexmedetomine group)

SUMMARY:
Anesthetic inhalation induction could be one of the most stressful experiences for children during the perioperative period, with almost 50% of them showing anxiety. It is an essential challenge for pediatric anesthesiologists on how to decrease anxiety for children in the operating room (OR) environment and to facilitate a smooth induction of anesthesia. Various factors like parental separation, unfamiliar surroundings, fear of physicians and needle injections can increase their preoperative anxiety. The researchers conducted the current study to investigate whether intranasal remimazolam can reduce anxiety in children before surgery.

DETAILED DESCRIPTION:
children aged 2-5 years old were randomly allocated into three equal groups based on the premedication routes: Group R with intranasal remimazolam, Group D with intranasal dexmedetomidine and Group P with intranasal placebo, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. with American Society of Anesthesiologists (ASA) physical status I or II；
2. aged 2-5 years；
3. children with weight for age within the normal range
4. were scheduled surgery with general anesthesia

Exclusion Criteria:

1. Children who had gastrointestinal,Cardiovascular or endocrine dysfunction;
2. contraindication to preoperative sedation or had a known allergy or hypersensitive reaction to either dexmedetomidine or remimazolam;
3. with any nasal pathology,organ dysfunction;
4. recently respiratory infection, mental disorder;
5. other reasons that researchers hold it is not appropriate to participate in this trial.-

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The level of anxiety | up to 30 minutes after study drug given
  The Modified Yale Preoperative Anxiety Scale:
  The 22-item measure has five behavioural categories: activity, emotional expressivity, alertness and arousal, vocalizations, and interaction with parents. Total scores range from 23.33 through 100 with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
The level of sedation | up to 30 minutes after study drug given
  Ramsay score
  1. Patient anxious or agitated or both
  2. Patient cooperative, oriented and tranquil
  3. Patient responds to commands only
  4. A brisk response to a light glabellar tap
  5. A sluggish response to a light glabellar tap
  6. No response higher scores mean a higher levels of sedation.
the compliance of study drug given | up to 30 minutes before anesthesia induction
  behavior score
  1. Clam and cooperative；
  2. Anxious but reassurable;
  3. Anxious but not reassurable;
  4. Crying, or resisting The scores of 1 and 2 signified satisfactory compliance, whereas scores of 3 and 4 were classified as poor compliance.
Parental separation anxiety scale | up to 30 minutes after study drug given
  A four-point parental separation anxiety scale as follows:
  1. Easy separation,
  2. Whimpers, but is easily reassured, not clinging,
  3. Cries and cannot be easily reassured, but not clinging to parents,
  4. Crying and clinging to parents. The scores of 1 and 2 signified acceptable separation whereas scores of 3 and 4 were classified as difficult separation.
The degree of cooperation during inhalation anesthesia induction | intraoperative, (During inhalation anesthesia induction)
  Induction Compliance Checklist range from 0 through 10,and lower scores indicate the higher degree of cooperation during inhalation anesthesia induction
Mask acceptance scale，MAS | intraoperative, (During inhalation anesthesia induction)
  Mask acceptance scale，MAS
  1. terrified, crying, agitated
  2. moderate fear, not calmed with reassurance
  3. slight fear of mask, easily calmed
  4. unafraid, cooperative, accepts mask readily The scores of 3 and 4 signified satisfactory mask acceptable whereas scores of 1 and 2 were classified as poor mask acceptable.
Pediatric anesthesia emergence delirium scale，PAEDs | Within up to 15-30 minutes after child's first eye opening in the postoperative period
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.pediatric anesthesia emergence delirium scale ≥12 at any time indicates presence of emergence delirium.
Recovery times | Within up to 30 minutes after child's first eye opening in the postoperative period
  The time from discontinuation of sevoflurane to the first open eye of the children and to achieve aldrete≥9
Number of children with adverse effects | Up to 24 hours including preoperative, intraoperative, and postoperative periods
  Number of children with adverse effects
  1. Bradycardia and/or hypotension need for hemodynamic support
  2. Desaturation is defined as Oxygen desaturation <90%
  3. Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Study Chair — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai YH, Wang CY, Fang YB, Ma HY, Gao YQ, Wang Z, Wu J, Lin H, Liu HC. Preoperative Anxiolytic and Sedative Effects of Intranasal Remimazolam and Dexmedetomidine: A Randomized Controlled Clinical Study in Children Undergoing General Surgeries. Drug Des Devel Ther. 2024 May 17;18:1613-1625. doi: 10.2147/DDDT.S461122. eCollection 2024. PMID 38774484